CLINICAL TRIAL: NCT01815944
Title: Onset Time of Brachial Plexus Block Using Local Anaesthetic Diluted With 0.9% Saline vs 5% Dextrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Mohd Shahnaz, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMMC883.11
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Comparison of Onset Time
Keywords: onset time; ultrasound-guided supraclavicular block; ropivacaine; normal saline; dextrose 5%
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.75% Ropivacaine and normal saline (Active Comparator): Ultrasound-guided supraclavicular block using 0.75% ropivacaine diluted with normal saline
  Interventions: Drug: 0.75% Ropivacaine; Drug: Normal saline
- 0.75% ropivacaine and dextrose 5% (Experimental): Ultrasound guided supraclavicular block using 0.75% ropivacaine diluted with dextrose 5%
  Interventions: Drug: 0.75% Ropivacaine; Drug: Dextrose 5%

INTERVENTIONS:
Drug: 0.75% Ropivacaine
  Other Names: Naropin
Drug: Normal saline
  Arms: 0.75% Ropivacaine and normal saline
Drug: Dextrose 5%
  Arms: 0.75% ropivacaine and dextrose 5%

SUMMARY:
Regional anesthesia employs the use of local anesthetics (LA) to block specific nerves to enable pain free surgery to be performed, or for intra and post operative pain relief. Dilution of local anesthetics with normal saline (NS) is a common practice to enable larger volumes of LA to be given, for example, in instances where multiple nerve blocks are needed to be performed for optimal pain relief while avoiding toxic doses.

A high sodium concentration is known to antagonize the analgesic effect of local anesthetics. 5% dextrose (D5W) on the other hand is painless on injection and does not cause any long-term effects in animals or humans when injected around neurological tissue. In the literature, only one study using dextrose 5% as diluent to produce 0.5% ropivacaine for axillary brachial plexus block showed a statistically significant reduction in the onset time for sensory blockade when compared with dilution with NS.

In this study, 0.5% ropivacaine diluted with D5W or NS is used for ultrasound guided supraclavicular brachial plexus block, and the time for complete sensory and motor blockade was compared. 0.5% ropivacaine is easily diluted and is a common concentration used at our centre for nerve blocks. The aim of this study is to assess if 0.5% ropivacaine diluted with D5W results in a shorter onset time for sensory block which may change the current practice of dilution with NS

DETAILED DESCRIPTION:
* Patients randomly assigned to receive either 0.5% ropivacaine diluted with NS or D5W.
* Randomization followed a computer-generated randomization table and patients are blinded as to their group allocation.
* Group allocations are concealed in a sealed opaque envelope and only known to an independent anaesthesia trainee who prepares 20mls 0.5% ropivacaine
* The anaesthesiologist involved in the performance of the supraclavicular brachial plexus block is blinded to group allocation
* All ultrasound-guided supraclavicular blocks are performed by 2 anaesthesiologists who are familiar with the technique.
* A trained anaesthesiology trainee who is blinded to group allocation evaluated sensory loss and motor blockade every 5 mins after injection of local anaesthetic.
* The extent of sensory loss is tested in the median, radial, ulnar, and musculocutaneous nerve distributions and evaluated using a 3-point score: 2 = normal sensation, 1 =loss of sensation to pinprick (ie, analgesia), or 0 = loss of sensation to light touch (ie, anesthesia). The extent of motor blockade is tested in the distribution of the radial (thumb abduction), ulnar (thumb adduction), musculocutaneous (flexion of the elbow in supination and pronation), and median nerves (thumb opposition) and evaluated using a 3-point scale where 2 = normal movement, 1 = paresis, and 0 = absent movement.
* Block success is defined as loss of sensation to pinprick (sensory score 1) in each of the radial, ulnar, median, and musculocutaneous nerve distributions measured 60 mins after the end of local anaesthetic injection. Patients in whom block success was not achieved after 60 mins were excluded from data analysis.
* During the postoperative recovery period, pain (verbal response score 4 or patient request for analgesic) is treated with IV tramadol 25-50 mg slow bolus with or without fentanyl 25mcg boluses every 5 minutes as needed.
* When oral intake is allowed, patients will receive oral paracetamol 1g with oral diclofenac 50 mg or celecoxib 200mg, if not contraindicated.
* The block duration is subsequently taken as time from complete analgesia to the time when the patient first feels the slightest pain from the operative site.
* Patients are followed up twice; once on post-operative day (POD) 1 and once between POD 7-10.
* They are seen in the ward or are contacted via telephone and asked for the presence of any pain, weakness, numbness, tingling, or any abnormal sensation in the operative extremity.
* If indicated, they are then told to come to hospital for further evaluation and management as necessary.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* elective or emergency surgery of the hand, forearm and elbow

Exclusion Criteria:

* diabetes mellitus
* neurological deficit
* contraindications to supraclavicular brachial plexus blockade
* unable to give consent
* patient refusal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Onset time for sensory blockade | 60 minutes

SECONDARY OUTCOMES:
Duration of sensory blockade | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: M. Shahnaz Hasan, MBBS, M Anes, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia